CLINICAL TRIAL: NCT07201636
Title: A Monocentre, Prospective, Longitudinal and Observational Natural History Study for Patients With Nemaline Myopathy
Brief Title: Natural History Study for Patients With Nemaline Myopathy in Belgium
Acronym: Acti-Nemaline
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Liege (Other)
Collaborators: Centre Hospitalier Régional de la Citadelle (Other); SYSNAV (Industry)
Responsible Party: Principal Investigator, Manon HUSTINX, Principal Investigator, Neurologist, Centre Hospitalier Universitaire de Liege
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Acti-Nemaline
Record Dates: First submitted 2025-08-21; First posted 2025-10-01 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Nemaline Myopathy
MeSH Terms: conditions — Myopathies, Nemaline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants with nemaline myopathy (Experimental)
  Interventions: Diagnostic Test: Motor Function Assessments; Device: Syde; Diagnostic Test: Respiratory Assessments; Diagnostic Test: Bulbar Function Questionnaires; Diagnostic Test: Clinical Global Impression (CGI); Other: Quality of Life Questionnaires; Procedure: Blood Sample Collection

INTERVENTIONS:
Diagnostic Test: Motor Function Assessments — The planned functional motor assessments are specific to age and degree of motor impairment. Participants are expected to have varying degrees of motor impairment, for example some will be non-ambulant. There is also a wide range of ages of participants. Therefore, some assessments will not be applicable. Some participants may gain or lose these abilities during the study and the assessments they complete shall be tailored accordingly aiming to reflect their most typical abilities on the day assessed.
Device: Syde — Syde is an innovative device intended to be used in a home-based environment. It is composed of two watch-like sensors, each containing a magneto-inertial sensors that record the linear acceleration, the angular velocity, the magnetic field of the movement in all directions.The two watches can be worn as wristwatch or placed near the ankle.
Diagnostic Test: Respiratory Assessments — The planned respiratory assessments are tailored to the participant's age and respiratory capacity. Participants are expected to have varying degrees of respiratory impairment, and some assessments may not be applicable to all. As participants may gain or lose respiratory function over the course of the study, the assessments completed will be adapted accordingly to reflect their most typical respiratory abilities on the day of assessment.
Diagnostic Test: Bulbar Function Questionnaires — The planned bulbar function assessments are age-specific and designed to reflect the participant's typical oral intake abilities. For participants aged 1-17 years, the Children's Eating and Drinking Activity Scale (CEDAS), will be used. For those aged 18 years and older, the Functional Oral Intake Scale (FOIS) will be applied. Both tools are part of a unified 7-item scale validated across paediatric and adult populations, ensuring continuity across age groups.
Diagnostic Test: Clinical Global Impression (CGI) — The Clinical Global Impression (CGI) tool will be used to assess overall disease severity and improvement across three functional domains: Physical Motor Function, Respiratory Function, and Bulbar Function. Assessments are based on clinician judgment using all available clinical data and are conducted by clinicians experienced with the disease under study.
Other: Quality of Life Questionnaires — The planned quality of life and functional status assessments are designed to capture the participant's overall well-being and daily functioning, taking into account the wide range of ages and disease severities in the study population. Validated questionnaires appropriate to age and functional level will be used to evaluate aspects such as health-related quality of life, fatigue, and daily activity limitations.
Procedure: Blood Sample Collection — Blood sample collection is usually done annually for NM patients as part of their standard of care. This is usually done by a nurse or a medical doctor according to standard guidelines for blood sampling. During routine blood sampling, additional blood will be collected and up to 20 ml of blood will be taken.

SUMMARY:
This is a prospective, longitudinal, observational study designed to characterize the natural history of Nemaline Myopathy (NM), a rare congenital neuromuscular disorder. The study will follow up to 10 participants of any age with genetically confirmed NM over a period of three years. Data will be collected during routine annual hospital visits and include clinical, motor, respiratory, and quality-of-life assessments. The goal is to improve clinical trial readiness by identifying disease-specific outcome measures and potential biomarkers.

DETAILED DESCRIPTION:
Nemaline Myopathies (NM) are a group of rare, genetically and clinically heterogeneous congenital myopathies characterized by the presence of nemaline bodies (rods) on muscle biopsy. The estimated incidence is approximately 1 in 50,000, though this is likely underestimated due to phenotypic variability and underdiagnosis of milder forms. NM typically presents in childhood, but adult-onset cases have been reported, often with retrospectively recognized early symptoms. Clinical manifestations range from severe neonatal presentations requiring mechanical ventilation, to milder forms compatible with ambulation and normal lifespan. Common features include congenital hypotonia, bulbar and respiratory involvement, and proximal muscle weakness, with sparing of extraocular muscles.

NM is associated with mutations in at least 12 genes, including NEB and ACTA1, which account for the majority of genetically confirmed cases. Inheritance patterns can be autosomal dominant or recessive. Despite advances in genetic diagnostics, a subset of patients remains without a confirmed molecular diagnosis.

Currently, treatment is supportive and aligned with general standards of care for congenital myopathies. However, several therapeutic strategies are in preclinical development, targeting gene-specific mechanisms, muscle function, and myogenesis. Clinical translation is challenged by disease rarity, heterogeneity, and the lack of validated outcome measures and biomarkers.

This monocentric study aims to address these gaps by prospectively observing up to 10 patients with NM over three years. Study assessments will coincide with routine annual hospital visits to minimize participant burden. For participants under 18 years of age, additional assessments at 6 and 18 months will be conducted to capture developmental changes.

Data collection will include:

Medical and neurological examinations Age- and ability-adapted motor and respiratory outcome measures Questionnaires assessing swallowing, fatigue, quality of life, and health economics.

Visit durations will vary based on age and ability, including standard care appointments. This study will provide critical longitudinal data to support the development of future clinical trials by identifying relevant outcome measures and potential biomarkers for NM.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* Any age
* Patient and/or parent or legal guardian must be willing and have the ability to provide written informed consent for participation in the study.
* Diagnosis of NM which in most cases includes having a disease-causing variant/s in one of the known NM causative genes and a consistent clinical phenotype.

Exclusion Criteria:

* Any confirmed chronic or acute condition or disease affecting any system(s), which could interfere with the results of the study and/or the compliance with the study procedures. This will be subject to the clinical judgement of the Coordinating Investigator (CI) and/or the Principal Investigator (PI).
* Clinically significant medical finding on the physical examination other than NM that, in the judgment of the Investigator, will make the patient unsuitable for participation in, and/or completion of the study procedures.
* Participants of ongoing (interventional) clinical trials that assess the efficacy of potential treatments will be excluded as assessments need to be done on the basis that represent the natural progression of NM.
* Safety concerns. This includes anything that might put the participant and/or their Parent(s) or Guardian(s) at risk through participating in the study potentially including but not limited to: Safeguarding concerns, Social Issues and Health issues.
* Ongoing pregnancy (for participants becoming pregnant during the trial, some assessments may be cancelled or postponed. This will be subject to the clinical judgement of the Coordinating Investigator and/or the Principal Investigator)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2029-04 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Change in Motor Function Measure (MFM32) Score | Over 3 years
  Difference in MFM32 score from baseline to each follow-up visit. The MFM32 is a validated scale (range 0-96; higher scores indicate better motor function).
Change in Ventilation Hours per Day | Over 3 years
  Evolution of the number of hours of assisted ventilation per day compared to baseline.

SECONDARY OUTCOMES:
Change in Quality of Life Score (PROMIS-29 Profile v2.1) | Over 3 years
  Difference in PROMIS-29 Profile v2.1 score from baseline to follow-up visits. PROMIS-29 includes 29 items across 7 domains (physical function, anxiety, depression, fatigue, sleep disturbance, social roles, pain interference) plus pain intensity. Higher T-scores indicate more of the concept being measured (e.g., higher fatigue score = more fatigue).
Drop-out Rate | Over 3 years
  Percentage of participants who discontinue participation before study completion.

OTHER OUTCOMES:
Change in Health Utilities Index 3 (HUI3) Score | Over 3 years
  Difference in HUI3 score from baseline to follow-up visits (range -0.36 to 1.00; higher scores indicate better health status).
Distance Walked per Hour | 6 recording periods of 1 month over 3 years
  Average distance walked per hour measured by wearable sensors.
Stride Speed Variability | 6 recording periods of 1 month over 3 years
  Coefficient of variation of stride speed measured by wearable sensors.
Number of Falls | 6 recording periods of 1 month over 3 years
  Number of falls recorded by wearable sensors during continuous monitoring in ambulant patients.

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Servais, MD, Study Director — Centre Hospitalier Universitaire de Liege
Locations (1):
- Centre de référence des maladies neuromusculaire, Centre Hospitalier Régional de la Citadelle, Liège, Belgium

IPD SHARING:
Plan to Share IPD: Undecided